CLINICAL TRIAL: NCT02948920
Title: Single Bolus Intravenous Ephedrine Attenuates Reduction of Core Body Temperature in Patients Undergoing Spinal Anesthesia for Arthroscopic Knee and Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Thanist Pravitharangul, MD, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-59-07; TCTR20161017007 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Body Temperature Changes
Keywords: ephedrine; core temperature; tympanic temperature; heat loss; spinal anesthesia; neuraxial; hypothermia; shivering
MeSH Terms: conditions — Body Temperature Changes; Hypothermia | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ephedrine (Experimental): Intravenous 9 mg of ephedrine (3 ml) given at finishing local anesthetic administration for spinal anesthesia
  Interventions: Drug: Ephedrine
- NSS (Placebo Comparator): Intravenous normal saline 3 ml given at finishing local anesthetic administration for spinal anesthesia
  Interventions: Drug: NSS

INTERVENTIONS:
Drug: Ephedrine — 9 mg of ephedrine (3 ml)
  Other Names: Experimental
  Arms: Ephedrine
Drug: NSS — 3 ml of normal saline
  Other Names: Control
  Arms: NSS

SUMMARY:
A prospective double-blinded randomized controlled study to determine efficacy of ephedrine in preserving core temperature in patients under neuraxial spinal anesthesia for knee and ankle arthroscopic surgery.

DETAILED DESCRIPTION:
To determine the effect of ephedrine on preserving core temperature (tympanic) when given at finishing of local anesthetic administration for spinal neuraxial anesthesia comparing to normal saline (120 minutes period)

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing knee or ankle arthroscopic surgery under spinal block at department of orthopaedic Ramathibodi Hospital
* BMI 17-30 kg/m2
* ASA physical status 1-3
* Age 18-70
* Last oral intake more than 6 hours (2 hours for water)
* Consent form acquired

Exclusion Criteria:

* Patient who are contraindicated for spinal block
* Anesthesia level higher than T4 or lower than T10
* Tympanic temperature more than 37.5 or less than 35.5 degrees Celsius
* Otitis or other ear infection
* Patients who receive alpha adrenergic blocker or beta adrenergic blocker
* Initial blood pressure presenting in operating theater 140 90 mmHg repeat after rest 5 minutes
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Tympanic temperature | 120 minutes
  Diffference of changes in tympanic membrane temperature at time points compare with baseline (before spinal block) between two groups

SECONDARY OUTCOMES:
Blood pressure | 120 minutes
  Difference of changes of blood pressure at time points compare with baseline (before spinal block) between two groups
Shivering | 120 minutes
  After performing spinal anesthesia in 120 minutes duration

CONTACTS AND LOCATIONS:
Overall Officials: Thanist Pravitharangul, MD, Principal Investigator — Department of Anesthesiology, Ramathibodi Hospital
Locations (1):
- Department of Anesthesiology, Ramathibodi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thanist Pravitharangul, Wirakorn Koopinpaitoon, Rungruedee Kraisen, Rojnarin Komonhirun. Ephedrine and propofol for induction of general anesthesia can decrease intraoperative hypothermia in patients undergoing plastic and breast surgery: a randomized, controlled trial. Asian Biomedicine Vol. 9 No. 3 June 2015; 379 - 385